CLINICAL TRIAL: NCT01103778
Title: Velcade Therapy for Severe IgA Nephropathy
Brief Title: Pilot Study of Velcade® in IgA Nephropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Rogosin Institute (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X05320; 1001010854 (Other: Weill Cornell Medical College IRB)
Record Dates: First submitted 2010-04-13; First posted 2010-04-15 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-10

CONDITIONS: Chronic Kidney Disease; IgA Nephropathy
Keywords: Chronic kidney disease; IgA nephropathy; Velcade®; Proteinuria; Bortezomib; Proteasome inhibitor
MeSH Terms: conditions — Renal Insufficiency, Chronic; Glomerulonephritis, IGA; Proteinuria | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Velcade® therapy (Experimental): Patients with greater than 1gm of proteinuria per day will receive Velcade®.
  Interventions: Drug: Bortezomib (Velcade®)

INTERVENTIONS:
Drug: Bortezomib (Velcade®) — Velcade® at 1.3 mg/m2, on days 1, 4, 8 and 11 (=1 cycle).
  Other Names: Velcade®; Bortezomib

SUMMARY:
The primary objective of this study is to investigate the ability of Velcade® (bortezomib) to induce complete or partial remission in patients with severe IgA nephropathy.

The secondary objectives are to assess clinical outcomes relating to safety and efficacy, such as infection, malignancy, preservation of renal function, partial responders, relapse rate, and to study mechanistic assays to predict remission.

DETAILED DESCRIPTION:
This exploratory single center, open-label, single treatment group assignment, safety and efficacy study will enroll 15 patients with severe IgA nephropathy. Subjects will receive 1 cycle of Velcade® to induce clinical remission. Follow-up visits will occur monthly for a year.

For this pilot study, the proportion of patients with clinical remission or partial response will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age or older.
2. Must have IgA nephropathy documented by kidney biopsy.
3. Must have greater than 1gm of proteinuria a day.
4. Must be on a stable dose of Angiotensin Converting Enzyme Inhibitor (ACEI) and/or Angiotensin Receptor Blocking agent (ARB) for at least 4 weeks prior to screening.

Exclusion Criteria:

1. Low platelet count and neutrophil count within certain limits defined for enrollment.
2. Underlying peripheral neuropathy.
3. Having cardiac problems, such as myocardial infarction, heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
4. Allergic to VELCADE®, boron or mannitol.
5. Female subjects who are pregnant or breast-feeding.
6. Recent use of investigational drug within 14 days before enrollment.
7. Having serious medical conditions and infections (including HIV,or hepatitis B or C) or psychiatric illness likely to interfere with participation in the study.
8. Diagnosed or treated for cancer within 3 years of participation in the study, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, and in situ malignancy, or low-risk prostate cancer after curative therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-07; Primary Completion 2017-04-17 (Actual); Study Completion 2017-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Choli Hartono, MD, Principal Investigator — The Rogosin Institute
Locations (1):
- The Rogosin Institute, New York, New York, United States

REFERENCES:
- [Result] Hartono C, Chung M, Perlman AS, Chevalier JM, Serur D, Seshan SV, Muthukumar T. Bortezomib for Reduction of Proteinuria in IgA Nephropathy. Kidney Int Rep. 2018 Mar 11;3(4):861-866. doi: 10.1016/j.ekir.2018.03.001. eCollection 2018 Jul. PMID 29988921
- [Derived] Yeo SC, Liew A, Barratt J. Emerging therapies in immunoglobulin A nephropathy. Nephrology (Carlton). 2015 Nov;20(11):788-800. doi: 10.1111/nep.12527. PMID 26032537
- [Derived] Hartono C, Muthukumar T. Treating IgA nephropathy: quid novi? Discov Med. 2014 Mar;17(93):131-8. PMID 24641955
- See also: The Rogosin Institute — http://www.rogosin.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Velcade Arm: Single treatment arm:
  Velcade® at 1.3 mg/m2, on days 1, 4, 8 and 11 (=1 cycle).
Period: Overall Study
Arm/Group | Velcade Arm
Started | 11
Completed | 8
Not Completed | 3
Not completed — Lost to Follow-up | 1
Not completed — Proteinuria improved prior to enrollment | 1
Not completed — Screen failure | 1

BASELINE CHARACTERISTICS:
Population: Patients with greater than 1gm of proteinuria per day will receive Velcade®.
Arm/Group | Velcade® Therapy
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 35 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Proteinuria
Description: Quantification of urinary protein will be made after treatment by measuring 24 hr urine protein.
Time Frame: Baseline and 1 year
Population: 1 participant was lost to followup.
Measure: Median (Full Range); unit: grams per 24 hrs
Arm/Group | Velcade® Therapy
Number analyzed (Participants) | 7
grams per 24 hrs
  Baseline | 2.52 [1.17 to 4.96]
  1 year | 1.43 [0.10 to 4.23]

2. Primary Outcome: Number of Participants With Complete Remission, Partial Response, or no Response.
Description: Complete remission was defined as daily proteinuria of less than 300mg measured by 24 hr urine collection.
  Partial response was defined as any reduction in daily proteinuria from baseline as measure by 24 hr urine collection.
Time Frame: 1 year
Population: 1 participant was lost to followup.
Measure: Count of Participants; unit: Participants
Arm/Group | Velcade Arm
Number analyzed (Participants) | 7
Participants
  Complete Remission | 3
  Partial Response | 1
  No Response | 3

3. Secondary Outcome: Serum Creatinine
Description: Preservation of renal function will be assessed.
Time Frame: Baseline and 1 year
Population: 1 participant lost to followup.
Measure: Median (Full Range); unit: milligram per deciliter
Groups:
- Velcade Arm: Single treatment arm
Arm/Group | Velcade Arm
Number analyzed (Participants) | 7
milligram per deciliter
  Baseline | 1.35 [0.54 to 2.63]
  1 year | 1.52 [0.52 to 2.75]

4. Secondary Outcome: Number of Participants With Abnormal Lab Values or Infections Related to Exposure to Study Medication.
Description: Complete blood count will be checked at regular intervals to monitor for anemia; liver panel; serum immunoglobulin profile will also be followed.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Velcade Arm
Number analyzed (Participants) | 8
Participants | 1

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Velcade® Therapy
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velcade® Therapy (N=8)
Mild reversible decline platelet count (Blood and lymphatic system disorders) | 1 (1) — Related to exposure to study medication

LIMITATIONS AND CAVEATS:
Our pilot study has several significant limitations, including small sample size, no control group, and nonrandomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-11-28): https://cdn.clinicaltrials.gov/large-docs/78/NCT01103778/Prot_SAP_000.pdf